CLINICAL TRIAL: NCT04385745
Title: BIODEGRADATION OF POLYLACTIDE-CO-GLYCOLIDE INTRAMEDULLARY NAILS USED IN TREATMENT OF CHILDREN'S FOREARM SHAFT FRACTURES AND CLINICAL RECOVERY OF THE PATIENTS IN THE LONG-TERM.
Brief Title: Treatment of Children's Forearm Shaft Fractures With Biodegradable Intramedullary Nailing, Compared With Elastic Stable Intramedullary Nailing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oulu University Hospital (Other)
Collaborators: Kanta-Häme Central Hospital (Other Government); Bioretec Ltd. (Industry)
Responsible Party: Principal Investigator, Jaakko Sinikumpu, Adjunct Professor, MD, PhD, Oulu University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: University of Oulu
Record Dates: First submitted 2020-05-04; First posted 2020-05-13 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Fractures, Bone; Injury Arm
MeSH Terms: conditions — Fractures, Bone; Arm Injuries

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled clinical trial.
Masking Description: Masking not possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elastic Stable Intramedullary Nailing (Experimental): BIN (biodegradable intramedullary nailing) method will be compared with the ESIN (elastic stable intramedullary nailing)
  Interventions: Procedure: Biodegradable Intramedullary Nailing (BIN)
- Biodegradable intramedullary nailing (Experimental): BIN method will be compared with the ESIN.
  Interventions: Procedure: Biodegradable Intramedullary Nailing (BIN)

INTERVENTIONS:
Procedure: Biodegradable Intramedullary Nailing (BIN) — Unstable forearm shaft fractures are treated by the study method (BIN) or the control method (ESIN).
  Other Names: Elastic Stable Intramedullary Nailing (ESIN)

SUMMARY:
The study purpose is to investigate long-term biodegradation process of the polylactide-co-glycolide (PLGA) intramedullary nails, used in treating the forearm shaft fractures in children. The primary objective of the study is to determine the stage of biodegradation of the polylactide-co-glycolide intramedullary nails, compared with the time since operation.

Biodegradation is to be evaluated by using Magnetic Resonance Imaging (MRI). Potential adverse events, being related to the biodegradation process of the implant, will be recognized: fluid accumulation, sinus formation, osteolysis, swelling, cyst formation and other soft-tissue reactions in the surroundings of the former fracture will be evaluated.

Radiographic recovery at least 4 years after the implant operation is secondary aims of the study. Radiographic investigation (plain radiographs in lateral and anterior-posterior views) are taken to evaluate the signs of bone healing after the long-bone diaphysis fracture, including the resolution of the previous callus formation, tubularization of the long-bones around the previous fracture area and remodeling of the angular and rotational alignment.

Clinical recovery in the long-term (at least 4 years) is another secondary aim of the study.

Prospective observational study will be performed. The study population comprises all the cases who were participating in the previous RCT ("BIOABSORBABLE INTRAMEDULLARY NAIL FIXATION OF FOREARM FRACTURES IN CHILDREN") and were therefore treated by means of biodegradable intramedullary nailing in years 2010 to 2015 (N=16).

All these patients will be invited and at least 4-year follow-up visit is performed at out-hospital clinics in the study institutions and radiographs and MRI will be taken. Flynn's criteria, MAYO elbow performance score and mini-DASH will be used. Health-related quality of life is to be analysed by using Pediatric Quality of Life Inventory (PedsQL). Visual analogue scale will be used for determining residual pain. A comprehensive analysis concerning the radiographic bone healing, according to Lane-Sandhu -scoring is determined and biodegradation of the implants, including the tricalciumphosphate tip will be evaluated by using MRI.

Number of Patients: N=15

Diagnosis and Main Criteria for Inclusion and Exclusion:

The study cases of the previous original research, described above, will be used to comprise the study population of the current project. The subject and/or guardian are invited to the study by a postal letter and by a call in case of no show. A signed and dated informed consent is required upon the participation.

Costs: The patients are to be investigated for long-term recovery according to the normal treatment protocol and no extra costs are caused for the patients or the institutes. The reason for further long-term follow-up and further imaging at four years' mark is that the implants were still visible in the patients at their last follow-up visit in two years' mark, in the previous research that has been terminated.

Safety and ethical consideration:

There are no health-related issues in clinical investigation and MRI of the patients. The plain radiographs of the upper extremities predispose the participants to radiation, with equivalence to 1-2 days of background radiation (www.stuk.fi, radiation doses). However, radiographs are not taken of gravidae females.

The study causes burden for the participants due to follow-up visit. In case of children and adolescents, the parents' presence is appreciated. However, long-term follow-up is justified because of the history of several injury and invasive surgical treatment performed and in order to certain the final degradation of the used implant.

Statistical Methods:

The radiographic and clinical findings will be reported in descriptive means. The mean, range and standard deviation (SD) will be reported for the continous variables. The issues in the short-term recovery and the potential association between the short-term findings and long-term results are analysed by using the SND test for independent variables. Further, the association of the clinical findings and subjective symptoms with the degradation stage of the implants will be investigated. Other appropriate statistical methods may also be used. All P-values are two-tailed and the level of significance is set as <0.05.

DETAILED DESCRIPTION:
This is a prospective observational clinical study in two centers in Finland. The study cannot be executed in a blinded fashion, because all patients treated by the study method will be invited.

The study purpose is to investigate long-term biodegradation process of the polylactide-co-glycolide intramedullary nails, used in treating the forearm shaft fractures in children. It is aimed to determine the stage of biodegradation of the polylactide-co-glycolide intramedullary nails, compared with the time since operation and the potential complications and/or radiographic and clinical recovery at least 4 years after the implant implementation.

Close clinical recovery is another objective of the study.

Potential adverse events, being related to the biodegradation process of the implant, are to be evaluated: fluid accumulation, sinus formation, osteolysis, swelling, cyst formation. Further, the soft-tissue reaction in the surroundings of the former fracture will be evaluated.

Radiographic recovery will be be evaluated in means of plain radiograph investigation (plain radiographs in lateral and anterior-posterior views). The signs of bone healing after the long-bone diaphysis fracture, including the resolution of the previous callus formation, tubularization of the long-bones around the previous fracture area, remodeling of the angular and rotational alignment will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* • Patients who have participated in the previous study, concerning the surgical treatment of forearm shaft fracture and have been treated by biodegradable intramedullary nailing (BIN), using the polylactide-co-glycolide nails (ActivaNail).

Exclusion Criteria:

* • The cases that have primarily been enrolled but interrupted the first study because of new fracture and been therefore surgically fixed with traditional (metallic) implants will be excluded.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2019-01-05 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Biodegradation of the implants and remodeling. Visibility of the implant in imaging (MRI, magnetic resonance imaging) | at least 4 years.
  Implant biodegradation and the remodeling of the fractured bone are to be evaluated by using different imaging modalities to view the residual implant. The biodegradation and remodeling will be described qualitatively, by the radiologist.
Biodegradation of the implants and remodeling. Visibility of the implant in imaging (radiographs) | at least 4 years
  Implant biodegradation and the remodeling of the fractured bone are to be evaluated by using different imaging modalities to view the residual implant. The biodegradation and remodeling will be described qualitatively, by the radiologist.

SECONDARY OUTCOMES:
Clinical recovery (forearm rotation motions) | at least 4 years postinjury
  Forearm rotation motion in pronation and supination (in left and right, by using a goniometer)
Clinical recovery (elbow motion) | at least 4 years postinjury
  Elbow motion by measuring a goniometer in left and right sides
Clinical recovery (carrying angle) | at least 4 years postinjury
  Ulno-humeral angle in degrees in left and right upper extremities
Clinical recovery (grip strength) | at least 4 years postinjury
  Grip strength by measured with using a hydraulic dynamometer in left and right sides

CONTACTS AND LOCATIONS:
Locations (1):
- Oulu University Hospital and University of Oulu, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No
Not applicable: there is a commercial sponsor who provided the implants and the study data is available only by request.